CLINICAL TRIAL: NCT01205724
Title: A Multi-National, Open-Label, Dose Escalation Trial, Evaluating Safety and Pharmacokinetics of Intravenous Doses of NNC 0129-0000-1003 in Patients With Haemophilia A
Brief Title: Safety and Pharmacokinetics of NNC 0129-0000-1003 in Subjects With Haemophilia A
Acronym: pathfinder™1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7088-3776; 2010-018520-68 (EudraCT Number); U1111-1116-2043 (Other: WHO); JapicCTI-101293 (Other: JAPIC)
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: turoctocog alfa pegol
- B (Experimental)
  Interventions: Drug: turoctocog alfa pegol
- C (Experimental)
  Interventions: Drug: turoctocog alfa pegol

INTERVENTIONS:
Drug: turoctocog alfa pegol — Single dose (low) administered intravenously (into the vein)
  Other Names: NNC 0129-0000-1003
  Arms: A
Drug: turoctocog alfa pegol — Single dose (medium) administered intravenously (into the vein)
  Other Names: NNC 0129-0000-1003
  Arms: B
Drug: turoctocog alfa pegol — Single dose (high) administered intravenously (into the vein)
  Other Names: NNC 0129-0000-1003
  Arms: C

SUMMARY:
This trial is conducted globally. The aim of this clinical trial is to investigate the safety and pharmacokinetics (the determination of the concentration of the administered medication in blood over time) of NNC 0129-0000-1003 in previously treated subjects with severe haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A
* Body Mass Index (BMI) below 35 kg/m2
* History of a minimum 150 exposure days (EDs) to FVIII products (prophylaxis/prevention/surgery/on-demand)

Exclusion Criteria:

* Any history of FVIII inhibitors
* Surgery planned to occur during the trial
* Platelet count less than 50,000 platelets/microlitre (assessed by laboratory)
* Congenital or acquired coagulation disorders other than haemophilia A

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) reported after administration of trial product | up to four weeks after trial product administration

SECONDARY OUTCOMES:
Area under the curve (AUC), total clearance (CL), terminal half-life (T½), incremental recovery (first sample) | from 0 to 168 hours after trial product administration
Safety assessment including physical examination, vital signs, electrocardiogram (ECG) and clinical laboratory assessments | up to four weeks after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (17):
- United States (5):
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Houston, Texas
- Germany (3):
  - Novo Nordisk Investigational Site, Frankfurt/M.
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Hanover
- Italy (2):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Vicenza
- Japan (3):
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Nagoya-shi, Aichi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Novo Nordisk Investigational Site, Bornova-IZMIR, Turkey (Türkiye)
- United Kingdom (2):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester

REFERENCES:
- [Result] Tiede A, Brand B, Fischer R, Kavakli K, Lentz SR, Matsushita T, Rea C, Knobe K, Viuff D. Enhancing the pharmacokinetic properties of recombinant factor VIII: first-in-human trial of glycoPEGylated recombinant factor VIII in patients with hemophilia A. J Thromb Haemost. 2013 Apr;11(4):670-8. doi: 10.1111/jth.12161. PMID 23398640
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com